CLINICAL TRIAL: NCT01817582
Title: A Randomized, Multi-Center, Parallel-Group, Safety and Efficacy Study of Lotemax® Gel 0.5% and Restasis 0.05% for 12 Weeks in Subjects With Mild or Moderate Keratoconjunctivitis Sicca (Dry Eye Disease; DED)
Brief Title: Lotemax® Gel 0.5% and Restasis 0.05% in Participants With Mild or Moderate Keratoconjunctivitis Sicca (Dry Eye Disease)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Collaborators: Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 813
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Results first posted 2019-08-30 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Dry Eye Disease
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — Loteprednol Etabonate; Cyclosporins; Health Services Needs and Demand

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lotemax Gel 0.5% and Restasis 0.05% (Experimental): Participants will administer lotemax gel 0.5 % BID in both eyes (OU) for 2 weeks, then administer both lotemax gel 0.5% and restasis emulsion 0.05% BID OU for 2 weeks, then administer restasis emulsion 0.05% BID OU for 8 weeks. Participants will also receive preservative-free Soothe Lubricant Eye Drops as needed (up to 4 times per day).
  Interventions: Drug: Lotemax; Drug: Restasis; Drug: Soothe® Lubricant Eye Drops
- Lotemax Gel 0.5% (Experimental): Participants will administer lotemax gel 0.5% BID OU for 12 weeks. Participants will also receive preservative-free Soothe Lubricant Eye Drops as needed (up to 4 times per day).
  Interventions: Drug: Lotemax; Drug: Soothe® Lubricant Eye Drops
- Restasis 0.05% (Active Comparator): Participants will administer restasis emulsion 0.05% BID OU for 12 weeks. Participants will also receive preservative-free Soothe Lubricant Eye Drops as needed (up to 4 times per day).
  Interventions: Drug: Restasis; Drug: Soothe® Lubricant Eye Drops

INTERVENTIONS:
Drug: Lotemax — Lotemax gel will be administered as per the dose and schedule specified in the arms.
  Other Names: loteprednol etabonate ophthalmic gel 0.5%
  Arms: Lotemax Gel 0.5%; Lotemax Gel 0.5% and Restasis 0.05%
Drug: Restasis — Restasis emulsion will be administered as per the dose and schedule specified in the arms.
  Other Names: cyclosporine ophthalmic emulsion 0.05%
  Arms: Lotemax Gel 0.5% and Restasis 0.05%; Restasis 0.05%
Drug: Soothe® Lubricant Eye Drops
  Other Names: Soothe lubricant eye drops will be administered as needed.

SUMMARY:
This study is being conducted to investigate the safety, comfort, and tolerability of 3 treatments: loteprednol etabonate ophthalmic (Lotemax®) gel 0.5 percent (%) administered twice daily (BID) with or without cyclosporine ophthalmic emulsion (Restasis) 0.05% administered BID, and Restasis 0.05% treatment alone for 12 weeks and at a follow-up safety visit 1 week post-treatment. This study will also investigate the relative efficacy of Lotemax gel 0.5% administered BID with or without Restasis 0.05% treatment administered BID and of Restasis 0.05% treatment alone for the reduction of clinical signs or symptoms of keratoconjunctivitis sicca (DED) over the first 4 weeks of a 12-week treatment period and at the end of a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with or treated for keratoconjunctivitis sicca (DED) within 6 months prior to screening visit (Day -14).
* Have a baseline intraocular pressure (IOP) measurement of greater than or equal to (≥) 5 millimeters of mercury (mmHg) and less than or equal to (≤) 22 mmHg in each eye, with or without anti-glaucoma therapy.
* Have mild to moderate DED in 1 eye or both eyes at screening visit (Day -14) and randomization visit (Day 0).

Exclusion Criteria:

* Have a known hypersensitivity to corticosteroids, cyclosporine, fluorescein, lissamine green, topical anesthetic, or any component of either of the study drugs.
* Have severe DED.
* Have corneal erosive disease or other conditions suggestive of extensive damage of the cornea.
* Have a history of elevated IOP, a history of glaucoma, or IOP greater than (>) 22 mmHg in either eye at the screening visit (Day -14).
* Have had penetrating intraocular surgery in the past 12 months or require penetrating intraocular surgery during the study.
* Have had eyelid surgery within the 6 months prior to Visit 1 (Day -14) or have DED secondary to surgery.
* Have visible evidence of anterior lid Demodex spp. infection or infestation.
* Have had corneal refractive surgery or corneal transplantation.
* Have congenitally absent lacrimal or meibomian glands or have any obstructive disease of the lacrimal glands, sarcoidosis, or any other lacrimal gland deficiency.
* Have a diagnosis of on-going ocular infection, active anterior blepharitis, moderate to severe pinguecula, Stevens-Johnson syndrome, ocular cicatricial pemphigoid, significant conjunctival scarring, ocular chemical burn, or ocular neurotrophic keratitis.
* Have any serious systemic disease or uncontrolled medical condition that in the judgment of the investigator could confound study assessments or limit compliance.
* Have a history of ocular herpetic keratitis or have had active blepharitis in the 4 weeks prior to the first dose.
* Have had ocular surgery (including laser) within 6 months prior to the first Treatment Period, or plan or require ocular surgery during the study. Neodymiumdoped:yttrium aluminum garnet (Nd:YAG) laser posterior capsulotomy is allowed.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2014-01-10 (Actual); Study Completion 2014-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Harris, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Bausch & Lomb Incorporated, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 102 participants were randomized in 1:1:1 to lotemax gel 0.5% and restasis 0.05%, lotemax gel 0.5%, or restasis 0.05% treatment groups.
Groups:
- Lotemax Gel 0.5% and Restasis 0.05%: Participants administered lotemax gel (loteprednol etabonate ophthalmic gel) 0.5 percent (%) twice daily (BID) in both eyes (OU) for 2 weeks, then administered both lotemax gel 0.5% and restasis emulsion (cyclosporin ophthalmic emulsion) 0.05% BID OU for 2 weeks, then administered restasis emulsion 0.05% BID OU for 8 weeks. Participants also received preservative-free Soothe Lubricant Eye Drops as needed (up to 4 times per day).
- Lotemax Gel 0.5%: Participants administered lotemax gel 0.5% BID OU for 12 weeks. Participants also received preservative-free Soothe Lubricant Eye Drops as needed (up to 4 times per day).
- Restasis 0.05%: Participants administered restasis emulsion 0.05% BID OU for 12 weeks. Participants also received preservative-free Soothe Lubricant Eye Drops as needed (up to 4 times per day).
Period: Overall Study
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Started | 33 | 36 | 33
Received at Least 1 Dose of Study Drug | 33 | 36 | 33
Completed | 31 | 35 | 33
Not Completed | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Participant revealed masked treatment | 1 | 0 | 0
Not completed — Randomized but exclusion criteria met | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Lotemax Gel 0.5% and Restasis 0.05%: Participants administered lotemax gel 0.5% BID OU for 2 weeks, then administered both lotemax gel 0.5% and restasis emulsion 0.05% BID OU for 2 weeks, then administered restasis emulsion 0.05% BID OU for 8 weeks. Participants also received preservative-free Soothe Lubricant Eye Drops as needed (up to 4 times per day).
- Total: Total of all reporting groups
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05% | Total
Number analyzed (Participants) | 33 | 36 | 33 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (8.30) | 64.3 (9.10) | 61.6 (9.98) | 62.7 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 26 | 81
  Male | 8 | 6 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Corneal Total Fluorescein Staining Score at for the Study Eye at Week 4
Description: Fluorescein Corneal Staining indicates the damage to the corneal epithelium (corneal epitheliopathy). Punctate corneal staining with fluorescein was evaluated and graded according to the National Eye Institute (NEI) grading method. The cornea was divided into 5 regions: central, superior, inferior, nasal and temporal. Each of these 5 regions was graded from scores 0 to 3, where 0 indicated no staining (absent) and 3 maximal staining (severe damage). The total score was the sum of all these regions, ranged from 0 (absence of corneal epitheliopathy) to 15 (severe corneal epitheliopathy).
Time Frame: Baseline (Day 0), Week 4
Population: ITT population included all randomized participants. Missing data was imputed using mixed-effect model for repeated measures (MMRM) method. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 32 | 36 | 33
units on a scale | -1.3 (1.95) | -1.7 (2.89) | -1.3 (1.63)
Statistical Analysis 1: Comparison: Lotemax Gel 0.5% and Restasis 0.05% vs Lotemax Gel 0.5%; Analysis was performed using MMRM method; Test type: Other; p = 0.6199, Mixed Models Analysis — Threshold for significance at 0.05 level; Least square (LS) mean difference = 0.3, 95% CI 2-sided [-0.7 to 1.3]
Statistical Analysis 2: Comparison: Lotemax Gel 0.5% and Restasis 0.05% vs Restasis 0.05%; Analysis was performed using MMRM method; Test type: Other; p = 0.8070, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = 0.1, 95% CI 2-sided [-0.9 to 1.2]
Statistical Analysis 3: Comparison: Lotemax Gel 0.5% vs Restasis 0.05%; Analysis was performed using MMRM method; Test type: Other; p = 0.8068, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -0.1, 95% CI 2-sided [-1.1 to 0.9]

2. Primary Outcome: Change From Baseline in Mean Ocular Surface Disease Index (OSDI) Questionnaire Total Score at Week 4
Description: OSDI is a 12-item questionnaire developed to assess severity of DED. There are 3 question types: "Have you experienced any of following (light sensitivity, eye feel gritty, sore eyes, blurred vision, and poor vision) during last week?"(items 1-5); "Have problems with your eyes limited you in performing any of following (reading, driving at night, working with computer, and watching TV) during last week?" (items 6-9); and "Have your eyes felt uncomfortable in any of following situations (windy, low humidity, air conditioned) during the last week?" (items 10-12). Response of each of these questions were graded on a scale (that relate to the frequency of ocular surface disease effects) of 0 (none of the time) to 4 (all of the time).Total OSDI score was calculated using following formula: OSDI=([sum of scores for all questions answered] × 100)/([total number of questions answered] * 4). Total OSDI score ranged from 0 to 100, with higher scores representing greater disability.
Time Frame: Baseline, Week 4
Population: ITT population included all randomized participants. Missing data was imputed using MMRM method. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 32 | 36 | 33
units on a scale | -5.2 (12.84) | -1.3 (17.04) | -0.6 (14.09)
Statistical Analysis 1: Comparison: Lotemax Gel 0.5% and Restasis 0.05% vs Lotemax Gel 0.5%; Analysis was performed using MMRM method; Test type: Other; p = 0.2296, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -4.4, 95% CI 2-sided [-11.6 to 2.8]
Statistical Analysis 2: Comparison: Lotemax Gel 0.5% and Restasis 0.05% vs Restasis 0.05%; Analysis was performed using MMRM method; Test type: Other; p = 0.1890, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -4.9, 95% CI 2-sided [-12.3 to 2.5]
Statistical Analysis 3: Comparison: Lotemax Gel 0.5% vs Restasis 0.05%; Analysis was performed using MMRM method; Test type: Other; p = 0.8836, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -0.5, 95% CI 2-sided [-7.7 to 6.7]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 13
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
percentage of participants | 27.3 | 25.0 | 27.3

4. Primary Outcome: Mean Grade for Participant-Reported Post-Dosing Ocular Comfort Values
Description: Participants scored their degree of comfort with their assigned study drug on a 4-point scale (0-3 units) within 5 minutes after instillation of study drug. Comfort grade 0 indicated comfortable, discomfort absent; 1 indicated generally comfortable, mild discomfort; 2 indicated some discomfort but tolerable, moderate discomfort; 3 indicated severely uncomfortable or intolerable. The mean global ocular comfort grade was reported.
Time Frame: Week 12
Population: Safety population included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 31 | 34 | 33
units on a scale | 0.5 (0.63) | 0.6 (0.92) | 0.5 (0.87)

5. Secondary Outcome: Change From Baseline in Mean OSDI Questionnaire Total Score and Individual Question Scores at Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: ITT population included all randomized participants. Here, 'Number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
units on a scale
  Light sensitivity: Baseline | 1.5 (0.97) | 1.5 (1.11) | 1.4 (0.99)
  Light sensitivity: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Light sensitivity: Change at Week 12 | -0.2 (1.17) | -0.1 (1.14) | -0.2 (1.36)
  Gritty feel: Baseline | 1.5 (0.97) | 1.4 (1.03) | 1.2 (0.80)
  Gritty feel: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Gritty feel: Change at Week 12 | -0.5 (1.09) | -0.4 (1.14) | -0.2 (1.10)
  Painful or sore eyes: Baseline | 1.0 (0.81) | 0.8 (0.77) | 0.8 (0.87)
  Painful or sore eyes: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Painful or sore eyes: Change at Week 12 | -0.2 (1.15) | -0.3 (0.83) | -0.2 (0.71)
  Blurred vision: Baseline | 0.9 (0.79) | 0.7 (0.79) | 0.9 (0.83)
  Blurred vision: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Blurred vision: Change at Week 12 | -0.2 (0.88) | -0.1 (0.91) | -0.1 (0.89)
  Poor vision: Baseline | 0.8 (0.77) | 0.7 (0.79) | 0.5 (0.71)
  Poor vision: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Poor vision: Change at Week 12 | -0.1 (0.94) | 0.1 (0.82) | 0.1 (0.93)
  Problem in reading: Baseline | 0.7 (0.72) | 0.8 (0.75) | 0.9 (0.77)
  Problem in reading: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Problem in reading: Change at Week 12 | 0.0 (0.68) | 0.0 (0.82) | -0.2 (1.07)
  Problem in driving at night: Baseline: number analyzed (Participants) | 29 | 30 | 29
  Problem in driving at night: Baseline | 0.9 (0.84) | 1.3 (1.01) | 1.1 (1.07)
  Problem in driving at night: Change at Week 12: number analyzed (Participants) | 25 | 27 | 29
  Problem in driving at night: Change at Week 12 | -0.2 (1.11) | 0.0 (1.22) | -0.2 (1.05)
  Problem in working with computer: Baseline: number analyzed (Participants) | 31 | 31 | 28
  Problem in working with computer: Baseline | 0.9 (0.81) | 1.0 (1.02) | 0.9 (0.80)
  Problem in working with computer:Change at Week12: number analyzed (Participants) | 29 | 28 | 28
  Problem in working with computer:Change at Week12 | -0.1 (0.90) | -0.2 (0.83) | -0.2 (0.83)
  Problem in watching TV: Baseline: number analyzed (Participants) | 33 | 36 | 32
  Problem in watching TV: Baseline | 0.9 (0.60) | 1.0 (0.94) | 0.8 (0.78)
  Problem in watching TV: Change at Week 12: number analyzed (Participants) | 31 | 35 | 32
  Problem in watching TV: Change at Week 12 | -0.4 (0.75) | -0.1 (1.13) | 0.1 (0.91)
  Uncomfortable in windy conditions: Baseline: number analyzed (Participants) | 29 | 32 | 28
  Uncomfortable in windy conditions: Baseline | 1.3 (1.04) | 1.5 (1.16) | 1.4 (1.00)
  Uncomfortable in windy condition:Change at Week12: number analyzed (Participants) | 25 | 29 | 28
  Uncomfortable in windy condition:Change at Week12 | -0.2 (1.12) | 0.0 (1.18) | 0.0 (1.33)
  Uncomfortable in low humidity: Baseline: number analyzed (Participants) | 27 | 32 | 30
  Uncomfortable in low humidity: Baseline | 1.5 (1.12) | 1.4 (1.08) | 1.3 (0.88)
  Uncomfortable in low humidity: Change at Week 12: number analyzed (Participants) | 22 | 27 | 28
  Uncomfortable in low humidity: Change at Week 12 | -0.7 (1.21) | 0.2 (1.00) | 0.0 (1.32)
  Uncomfortable in air conditioning: Baseline: number analyzed (Participants) | 33 | 35 | 33
  Uncomfortable in air conditioning: Baseline | 1.5 (0.97) | 1.5 (1.07) | 1.6 (0.87)
  Uncomfortable in air conditioning:Change at Week12: number analyzed (Participants) | 21 | 26 | 26
  Uncomfortable in air conditioning:Change at Week12 | -0.3 (1.11) | -0.3 (1.43) | -0.8 (1.34)
  Total OSDI score: Baseline | 27.9 (8.41) | 27.8 (9.18) | 26.5 (8.12)
  Total OSDI score: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Total OSDI score: Change at Week 12 | -5.6 (14.50) | -3.2 (15.05) | -4.0 (15.14)

6. Secondary Outcome: Change From Baseline in Mean Corneal Total Fluorescein Staining Score for the Study Eye and Averaged for Both Eyes at Week 12
Description: Fluorescein Corneal Staining indicates the damage to the corneal epithelium (corneal epitheliopathy). Punctate corneal staining with fluorescein was evaluated and graded according to the NEI grading method. The cornea was divided into 5 regions: central, superior, inferior, nasal and temporal. Each of these 5 regions was graded from scores 0 to 3, where 0 indicated no staining (absent) and 3 maximal staining (severe damage). The total score was the sum of all these regions, ranged from 0 (absence of corneal epitheliopathy) to 15 (severe corneal epitheliopathy).
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
units on a scale
  Score for study eye: Baseline | 5.6 (1.92) | 5.7 (2.19) | 5.5 (1.97)
  Score for study eye: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Score for study eye: Change at Week 12 | -1.3 (2.30) | -0.7 (3.01) | -1.6 (2.46)
  Score for both eyes: Baseline | 5.02 (1.637) | 5.22 (1.955) | 5.08 (1.896)
  Score for both eyes: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Score for both eyes: Change at Week 12 | -0.66 (1.809) | -0.69 (2.400) | -1.17 (2.207)

7. Secondary Outcome: Change From Baseline in Mean Value of Participant Worst Eye Score for Each Symptom (Including the Pre-Specified Worst Symptom) in the List of Possible Worst Symptoms at Week 12
Description: Participants eligible for enrollment rated the severity of dry eye symptoms at Baseline (Day 0) on a 5-point grading scale (ranged from 0 [no problem] to 4 [continuous or severe discomfort; intolerable]) for each of 8 symptoms in the following symptom list prior to enrollment and then selected their most bothersome symptom: Photophobia, itchiness or scratchiness, grittiness or sandiness, foreign body sensation, haziness or blurriness, eye discomfort, burning or stinging, or photopsia (sensation of light or light flashes). Participants subsequently rated their dry eye symptom severity on the same 5-point grading scale at Week 2-Week 12 for study eye for the worst symptom identified at Baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
units on a scale
  Burning or stinging: Baseline | 1.2 (1.12) | 1.2 (1.28) | 1.0 (1.24)
  Burning or stinging: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Burning or stinging: Change at Week 12 | -0.5 (1.23) | -0.6 (1.26) | -0.3 (1.35)
  Eye discomfort: Baseline | 1.5 (1.03) | 1.8 (1.17) | 1.8 (1.06)
  Eye discomfort: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Eye discomfort: Change at Week 12 | -0.5 (1.26) | -0.9 (1.06) | -1.1 (0.97)
  Foreign body sensation: Baseline | 0.9 (0.98) | 1.3 (1.19) | 1.0 (0.95)
  Foreign body sensation: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Foreign body sensation: Change at Week 12 | -0.3 (1.40) | -0.6 (1.27) | -0.5 (1.03)
  Grittiness or sandiness: Baseline | 1.5 (1.15) | 1.6 (1.16) | 1.3 (1.05)
  Grittiness or sandiness: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Grittiness or sandiness: Change at Week 12 | -0.5 (1.18) | -0.8 (1.10) | -0.5 (1.39)
  Haziness or blurriness: Baseline | 1.2 (0.87) | 1.2 (1.12) | 1.3 (1.18)
  Haziness or blurriness: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Haziness or blurriness: Change at Week 12 | -0.4 (0.88) | -0.3 (1.24) | -0.6 (1.03)
  Itchiness or scratchiness: Baseline | 1.4 (0.99) | 1.5 (1.23) | 1.5 (0.97)
  Itchiness or scratchiness: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Itchiness or scratchiness: Change at Week 12 | -0.4 (1.28) | -0.6 (1.17) | -0.5 (1.12)
  Photophobia: Baseline | 1.3 (1.21) | 1.4 (1.23) | 1.5 (1.09)
  Photophobia: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Photophobia: Change at Week 12 | -0.2 (1.05) | -0.2 (1.21) | -0.5 (1.03)
  Photopsia: Baseline | 0.2 (0.46) | 0.3 (0.51) | 0.3 (0.85)
  Photopsia: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Photopsia: Change at Week 12 | 0.0 (0.66) | -0.1 (0.56) | -0.1 (1.10)
  Worst dry eye symptom: Baseline | 2.2 (0.96) | 2.6 (0.94) | 2.5 (0.94)
  Worst dry eye symptom: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Worst dry eye symptom: Change at Week 12 | -0.8 (1.34) | -1.3 (1.23) | -1.5 (1.12)

8. Secondary Outcome: Change From Baseline in Mean Total Combined Lissamine Green (LG) Staining (Nasal Plus Temporal Conjunctival) Score for the Study Eye and Averaged for Both Eyes at Week 12
Description: LG staining is useful for monitoring evidence of eye dryness in conjunctival tissue. Scoring of conjunctival staining was done using Oxford conjunctival grading scale. The investigator instilled an ophthalmic dye (LG stain) on the eye and rated staining in 2 areas (nasal and temporal conjunctiva). Staining was rated on a 6-point scale from 0 (absent) to 5 (severe). The total score ranged from 0 (improvement; no conjunctival damage) to 12 (worsening; severe conjunctival damage).
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
units on a scale
  Score for study eye: Baseline: number analyzed (Participants) | 31 | 36 | 32
  Score for study eye: Baseline | 8.5 (5.10) | 9.2 (4.68) | 7.7 (4.50)
  Score for study eye: Change at Week 12: number analyzed (Participants) | 29 | 34 | 32
  Score for study eye: Change at Week 12 | -0.9 (4.31) | -1.8 (5.45) | -1.2 (4.32)
  Score for both eyes: Baseline: number analyzed (Participants) | 31 | 36 | 32
  Score for both eyes: Baseline | 8.37 (5.045) | 9.06 (4.107) | 7.35 (4.542)
  Score for both eyes: Change at Week 12: number analyzed (Participants) | 29 | 34 | 32
  Score for both eyes: Change at Week 12 | -0.98 (4.195) | -1.82 (4.927) | -0.75 (4.811)

9. Secondary Outcome: Change From Baseline in Mean Tear Osmolarity of Participant Worst Eye Value at Week 12
Description: Tear osmolarity was measured with the TearLab Osmolarity System. The TearLab instrument measures the impedance of 50 nanoliters (nL) tear samples taken with a disposable lab-on-a-chip device. Tear samples from enrolled participants were taken at Weeks 2, 4, and 12 from each eye in duplicate with a tear sampler according to the manufacturer's instructions, and the tear osmolarity for each sample was read with the TearLab instrument. Osmolarity values were provided by the TearLab instrument in 3-digit units of milliosmoles (mOsm). Change from mean baseline values for all participants within a treatment group was calculated using a participant's worst eye value at Week 12.
Time Frame: Baseline, Week 12
Population: ITT population included all randomized participants. Here, 'Number analyzed' signifies participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: mOsm
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
mOsm
  Baseline: number analyzed (Participants) | 20 | 22 | 20
  Baseline | 312.1 (11.48) | 307.4 (8.91) | 311.6 (17.11)
  Change at Week 12: number analyzed (Participants) | 18 | 21 | 20
  Change at Week 12 | 0.7 (16.67) | 4.3 (9.88) | -1.5 (17.33)

10. Secondary Outcome: Change From Baseline in Mean Tear Osmolarity Between Two Eyes of Participant at Week 12
Description: Tear osmolarity was measured with the TearLab Osmolarity System. The TearLab instrument measures the impedance of 50 nL tear samples taken with a disposable lab-on-a-chip device. Tear samples from enrolled participants were taken at Weeks 2, 4, and 12 from each eye in duplicate with a tear sampler according to the manufacturer's instructions, and the tear osmolarity for each sample was read with the TearLab instrument. Osmolarity values were provided by the TearLab instrument in 3-digit units of mOsm. Change from mean baseline values for all participants within a treatment group was calculated for the difference between average values between 2 eyes at Week 12.
Time Frame: Baseline, Week 12
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mOsm
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
mOsm
  Baseline: number analyzed (Participants) | 20 | 22 | 20
  Baseline | 7.9 (5.72) | 5.4 (4.62) | 7.2 (10.44)
  Change at Week 12: number analyzed (Participants) | 18 | 21 | 20
  Change at Week 12 | 0.6 (9.70) | 2.9 (6.62) | -0.3 (11.52)

11. Secondary Outcome: Change From Baseline in Mean Eye Comfort Index Questionnaire Total Score and Individual Question Scores at Week 12
Description: An ocular comfort assessment questionnaire was administered at weeks 2, 4, and 12 to participants. The assessment of the degree of dry eye discomfort experienced by the participant was conducted using an adapted and validated 12-item ocular comfort questionnaire ( to measure the frequency and intensity of 6 common dry eye symptoms: dryness, grittiness, stinging, eye tiredness, pain, and itching) based upon the ocular comfort index of Johnson and Murphy. Each item (question) was graded from 0 to 4, where 0 = Not at all, 1 = Seldom; perceptible but not intense, 2 = Sometimes; intermittent with easily tolerable intensity, 3 = Frequently; often but with tolerable intensity, 4 = Constantly; constant or intolerable intensity. Total score was calculated and normalized to a score of 0 (no discomfort)-100 (more ocular discomfort) by the formula: Normalized comfort grade = ([Total Comfort Grade] * 100)/48.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
units on a scale
  Dryness: Baseline | 2.3 (0.85) | 2.2 (0.81) | 2.2 (0.93)
  Dryness: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Dryness: Change at Week 12 | -0.4 (0.92) | -0.1 (0.99) | -0.4 (0.87)
  Dryness intensity: Baseline | 2.2 (0.93) | 2.1 (0.90) | 2.2 (0.92)
  Dryness intensity: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Dryness intensity: Change at Week 12 | -0.5 (0.93) | -0.3 (1.06) | -0.6 (1.08)
  Grittiness: Baseline | 1.5 (0.90) | 1.7 (1.09) | 1.4 (0.97)
  Grittiness: Change at Week 12: number analyzed (Participants) | 30 | 34 | 33
  Grittiness: Change at Week 12 | -0.4 (0.97) | -0.6 (0.95) | -0.6 (1.06)
  Grittiness intensity: Baseline | 1.6 (1.06) | 1.6 (0.93) | 1.3 (0.98)
  Grittiness intensity: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Grittiness intensity: Change at Week 12 | -0.5 (0.96) | -0.6 (0.96) | -0.5 (1.03)
  Stinging: Baseline | 1.3 (1.07) | 1.2 (1.15) | 1.0 (0.79)
  Stinging: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Stinging: Change at Week 12 | -0.2 (1.17) | -0.4 (1.13) | -0.1 (1.38)
  Stinging intensity: Baseline | 1.2 (1.06) | 1.3 (1.16) | 1.0 (0.85)
  Stinging intensity: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Stinging intensity: Change at Week 12 | -0.2 (0.93) | -0.4 (1.11) | -0.1 (1.23)
  Tiredness: Baseline | 1.8 (1.01) | 1.6 (0.93) | 1.9 (1.02)
  Tiredness: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Tiredness: Change at Week 12 | -0.4 (1.11) | -0.2 (0.77) | -0.4 (0.83)
  Tiredness intensity: Baseline | 1.7 (1.02) | 1.6 (1.02) | 1.8 (1.00)
  Tiredness intensity: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Tiredness intensity: Change at Week 12 | -0.3 (1.03) | -0.2 (0.90) | -0.4 (0.70)
  Pain: Baseline | 0.9 (0.89) | 0.8 (0.81) | 0.7 (0.69)
  Pain: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Pain: Change at Week 12 | -0.2 (0.92) | -0.2 (0.96) | -0.2 (0.76)
  Pain intensity: Baseline | 0.9 (0.98) | 0.8 (0.97) | 0.8 (0.88)
  Pain intensity: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Pain intensity: Change at Week 12 | -0.1 (1.02) | -0.3 (1.07) | -0.3 (0.74)
  Itch: Baseline | 1.5 (1.03) | 1.6 (1.16) | 1.2 (0.99)
  Itch: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Itch: Change at Week 12 | -0.2 (1.34) | -0.7 (1.32) | -0.2 (1.07)
  Itch intensity: Baseline | 1.5 (1.03) | 1.5 (1.16) | 1.2 (1.09)
  Itch intensity: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Itch intensity: Change at Week 12 | -0.2 (1.19) | -0.7 (1.22) | -0.3 (1.10)
  Total comfort score: Baseline | 38.4 (16.39) | 37.8 (16.99) | 34.8 (14.06)
  Total comfort score: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Total comfort score: Change at Week 12 | -7.2 (17.16) | -10.0 (16.35) | -8.6 (14.48)

12. Secondary Outcome: Change From Baseline in Mean Eye Dryness Questionnaire Total and Individual Question Scores at Week 12
Description: The 5-item Dry Eye Questionnaire (DEQ-5) is a validated questionnaire for discriminating self-assessed severity of dry eye diagnoses. The participants rated the frequency on a scale of 0 (never) to 4 (constant) with which they have experienced 3 symptoms (watery eyes, discomfort and dryness). The participant was also asked to rate the increase in intensity of discomfort and dryness throughout the day on a scale of 0 (never have it) to 5 (very intense). Participant rated the overall severity of dry eye symptoms on a scale of 0 (no problem) to 4 (intolerable; unable to perform my daily tasks). Total DEQ-5 score was the sum of scores for frequency and intensity of dryness and discomfort plus frequency of watery eyes. A DEQ-5 total score >6 was indicative of DED and a score >12 is indicative of Sjögren's syndrome.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
units on a scale
  Discomfort frequency: Baseline | 2.2 (0.81) | 2.1 (0.67) | 2.1 (0.82)
  Discomfort frequency: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Discomfort frequency: Change at Week 12 | -0.4 (0.67) | -0.2 (0.97) | -0.3 (0.94)
  Discomfort intensity: Baseline | 2.4 (1.14) | 2.5 (1.03) | 2.4 (1.22)
  Discomfort intensity: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Discomfort intensity: Change at Week 12 | -0.4 (1.20) | -0.5 (0.85) | -0.4 (1.11)
  Dryness frequency: Baseline | 2.4 (0.79) | 2.1 (0.82) | 2.4 (1.00)
  Dryness frequency: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Dryness frequency: Change at Week 12 | -0.6 (0.80) | -0.1 (0.83) | -0.6 (1.00)
  Dryness intensity: Baseline | 2.4 (1.15) | 2.8 (1.08) | 2.3 (1.27)
  Dryness intensity: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Dryness intensity: Change at Week 12 | -0.2 (1.31) | -0.7 (0.83) | -0.4 (1.32)
  Watery eyes frequency: Baseline | 1.5 (1.00) | 1.3 (1.03) | 1.3 (1.16)
  Watery eyes frequency: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Watery eyes frequency: Change at Week 12 | -0.4 (1.14) | -0.4 (0.77) | 0.0 (1.37)
  Overall severity: Baseline | 1.9 (0.77) | 1.8 (0.82) | 1.8 (0.79)
  Overall severity: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Overall severity: Change at Week 12 | -0.6 (0.92) | -0.4 (0.97) | -0.5 (0.71)
  Total score: Baseline | 11.0 (3.60) | 10.8 (3.38) | 10.6 (4.55)
  Total score: Change at Week 12: number analyzed (Participants) | 31 | 35 | 33
  Total score: Change at Week 12 | -2.0 (3.52) | -2.0 (2.81) | -1.6 (4.08)

13. Secondary Outcome: Change From Baseline in Mean Tear Film Breakup Time (TFBUT) (by Fluorescein Staining) of the Study Eye and Averaged for Both Eyes of a Participant at Week 12
Description: The TFBUT was defined as the interval between the last complete blink and the first appearance of dark zones or spots, or disruption in the tear film. Tear film breakup time is a measure of the stability of the tear film protecting the cornea and bulbar conjunctiva. 5 microliters (μL) of fluorescein solution was instilled in the participant's eye, after which the participant blinked several times, then kept the eye open. The cornea was visualized through the slit lamp using appropriate barrier filters for the white light source.
  TFBUT was counted using a stopwatch. Three consecutive measurements were taken and averaged for actual TFBUT. TFBUT at Baseline (Day 0) was subtracted from TFBUT at Week 12 (Day 84) and reported as change. A higher number represented a lengthening in the TFBUT. A longer TFBUT indicated a more stable tear film.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
seconds
  Study eye: Baseline | 2.87 (1.715) | 3.23 (1.739) | 3.09 (1.546)
  Study eye: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Study eye: Change at Week 12 | 0.25 (2.106) | 0.32 (2.038) | 0.16 (1.807)
  Both eyes: Baseline | 3.01 (2.042) | 3.28 (1.902) | 3.45 (2.371)
  Both eyes: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Both eyes: Change at Week 12 | 0.17 (2.019) | 0.57 (2.305) | -0.17 (2.286)

14. Secondary Outcome: Change From Baseline in Mean Non-Invasive Keratographic Tear Film Breakup Time (NIKBUT) of the Study Eye and Averaged for Both Eyes of a Participant at Week 12
Description: The tear film breakup time was defined as the interval between the last complete blink and the first appearance of dark zones or spots, or disruption in the tear film. Tear film examination using any non-invasive method analyzes optical reflections from the cornea. Reflections that become distorted are characteristic of tear film breakup. Circular images were projected onto the corneal surface using an Oculus Keratograph 5M instrument, and the tear film reflection was observed on a computer. NIKBUT (initial break-up time [NIKBUTi] and average break-up time [NIKBUTav]) were determined and recorded for each eye in duplicate after participant blink 2 times. NIKBUT at Baseline (Day 0) was subtracted from NIKBUT at Week 12 (Day 84) and reported as change. A higher number represented a lengthening in the NIKBUT. A longer NIKBUT indicated a more stable tear film.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
seconds
  NIKBUTi for study eye: Baseline: number analyzed (Participants) | 10 | 13 | 12
  NIKBUTi for study eye: Baseline | 6.49 (1.349) | 8.11 (3.531) | 7.18 (4.867)
  NIKBUTi for study eye: Change at Week 12: number analyzed (Participants) | 9 | 12 | 11
  NIKBUTi for study eye: Change at Week 12 | 0.59 (3.826) | 1.09 (5.833) | 0.31 (6.356)
  NIKBUTi for both eyes: Baseline: number analyzed (Participants) | 10 | 13 | 13
  NIKBUTi for both eyes: Baseline | 6.92 (2.175) | 8.22 (4.240) | 7.60 (4.896)
  NIKBUTi for both eyes: Change at Wee 12: number analyzed (Participants) | 9 | 13 | 12
  NIKBUTi for both eyes: Change at Wee 12 | -0.14 (2.774) | 0.17 (3.511) | -1.08 (4.770)
  NIKBUTav for study eye: Baseline: number analyzed (Participants) | 10 | 13 | 12
  NIKBUTav for study eye: Baseline | 9.57 (3.018) | 11.20 (3.164) | 9.07 (5.595)
  NIKBUTav for study eye: Change at Week 12: number analyzed (Participants) | 9 | 12 | 11
  NIKBUTav for study eye: Change at Week 12 | -0.01 (2.806) | 1.55 (5.453) | 1.26 (5.636)
  NIKBUTav for both eyes: Baseline: number analyzed (Participants) | 10 | 13 | 13
  NIKBUTav for both eyes: Baseline | 9.21 (3.253) | 10.99 (3.969) | 9.98 (5.744)
  NIKBUTav for both eyes: Change at Week 12: number analyzed (Participants) | 9 | 13 | 12
  NIKBUTav for both eyes: Change at Week 12 | -0.04 (1.882) | 1.32 (3.985) | 0.04 (5.117)

15. Secondary Outcome: Change From Baseline in Mean Anesthetized Schirmer's Test Values (Distance of Strips Wetting) in the Study Eye and Averaged for Both Eyes of a Participant at Week 13
Description: Schirmer's test measures the aqueous component of tear secretion. The Schirmer's test (anesthetized) is a measure of the tonic secretion of the aqueous component of tears. A Schirmer's test (with anaesthesia) was performed for both eyes of a participant using Schirmer's test strips. After instillation of an ophthalmic anaesthetic, Schirmer's test strips for each eye were left in place for 5 minutes with participant eyelids closed. After 5 minutes, the Schirmer's test strips were removed with forceps and the distance to where each strip was wetted was recorded in millimeters (mm). Lesser wetting of strips (low levels of tear production) were associated with dry eye.
Time Frame: Baseline, Week 13
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
mm
  Wetting distance for Study eye: Baseline | 6.1 (1.89) | 6.6 (2.18) | 6.6 (2.08)
  Wetting distance for Study eye: Change at Week 13: number analyzed (Participants) | 31 | 35 | 33
  Wetting distance for Study eye: Change at Week 13 | 2.5 (6.16) | 1.7 (6.59) | 2.5 (5.55)
  Wetting distance for both eyes: Baseline | 6.66 (1.76) | 6.78 (2.01) | 6.76 (1.90)
  Wetting distance for both eyes: Change at Week 13: number analyzed (Participants) | 31 | 35 | 33
  Wetting distance for both eyes: Change at Week 13 | 2.17 (5.72) | 1.39 (5.61) | 2.59 (5.29)

16. Secondary Outcome: Averaged Daily Soothe Lubricant Eye Drops Usage
Description: Amount of averaged daily soothe lubricant eye drops (Bausch + Lomb) used was reported.
Time Frame: Baseline up to Week 12
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: drops/day
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
drops/day | 2.07 (1.013) | 1.79 (1.073) | 2.04 (1.075)

17. Secondary Outcome: Number of Participants With Overall Change From Baseline in Dry Symptoms at Week 12 as Assessed Independently by Investigators and Participants
Description: Participants and investigators independently rated the overall change from baseline in dry eye conditions for each participant on a 7-point Likert scale at Week 12. The scale ranged from +3 to -3, where +3 = Substantial improvement in dry eye; little or no awareness of dry eye, +2 = Some improvement in dry eye, +1 = Little improvement in dry eye, 0 = No improvement in dry eye, -1 = Slight worsening of dry eye, -2 = Some worsening of dry eye, and -3 = Substantial worsening of dry eye.
Time Frame: Baseline, Week 12
Population: ITT population included all randomized participants. Here, 'Overall number of participants analyzed' signifies participants evaluable for specified categories; that is, participants who had investigator global improvement assessment or participant-reported global improvement assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 31 | 34 | 33
Participants
  Investigator-reported:: +3 | 0 | 2 | 3
  Investigator-reported:: +2 | 7 | 11 | 10
  Investigator-reported:: +1 | 16 | 12 | 14
  Investigator-reported:: 0 | 5 | 8 | 4
  Investigator-reported:: -1 | 2 | 1 | 1
  Investigator-reported:: -2 | 1 | 0 | 1
  Investigator-reported:: -3 | 0 | 0 | 0
  Participant-reported:: +3 | 4 | 6 | 9
  Participant-reported:: +2 | 10 | 15 | 14
  Participant-reported:: +1 | 8 | 7 | 7
  Participant-reported:: 0 | 6 | 5 | 2
  Participant-reported:: -1 | 2 | 1 | 1
  Participant-reported:: -2 | 0 | 0 | 0
  Participant-reported:: -3 | 1 | 0 | 0

18. Secondary Outcome: Change From Baseline in Ocular Redness Score for Study Eye and Averaged for Both Eyes at Week 12, as Assessed by Investigator
Description: The Investigator subjectively rated the degree of eye redness on a 4-point (0-3) grading scale prior to any objective grading of eye redness for a participant, where score 0 = none absent; no redness present in the white of the eyes, 1 = mild, slightly dilated blood vessels seen in some portion of the white of the eyes; the color of vessels was typically pink, 2 = moderate more apparent dilation of blood vessels in the white of the eyes; vessel color was more intense (redder) and involves the majority of the vessel bed, 3 = severe numerous obvious dilated blood vessels throughout the white of the eyes; the vessel color was deep red.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
units on a scale
  Redness of study eye: Baseline | 1.0 (0.79) | 1.0 (0.70) | 1.0 (0.68)
  Redness of study eye: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Redness of study eye: Change at Week 12 | -0.1 (0.60) | -0.2 (0.69) | -0.1 (0.66)
  Redness of both eyes: Baseline | 1.00 (0.760) | 0.97 (0.696) | 1.06 (0.726)
  Redness of both eyes: Change at Week 12: number analyzed (Participants) | 31 | 34 | 33
  Redness of both eyes: Change at Week 12 | -0.10 (0.583) | -0.21 (0.698) | -0.12 (0.625)

19. Secondary Outcome: Change From Baseline in Non-Invasive Keratographic Limbal and Bulbar Ocular Redness Scores for Study Eye and Averaged for Both Eyes at Week 12, as Assessed by Investigator
Description: The objective redness scoring assessment was conducted by automated means using an Oculus Keratograph 5M. Duplicate digital photographs of bulbar and limbal conjunctiva were taken with the Oculus Keratograph 5M instrument for each eye of a participant and the images were analyzed using R-Scan classification software to numerically rate the severity of ocular redness (bulbar and limbal redness) on a 4-point (0-3) grading scale, where score 0 = none absent; no redness present in the white of the eyes, 1 = mild, slightly dilated blood vessels seen in some portion of white of the eyes; color of vessels was typically pink, 2 = moderate more apparent dilation of blood vessels in the white of the eyes; vessel color was more intense (redder) and involves the majority of the vessel bed, 3 = severe numerous obvious dilated blood vessels throughout the white of the eyes; the vessel color was deep red. Keratograph 5M ocular redness grading results were averaged for each eye and for both eyes.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Number analyzed (Participants) | 33 | 36 | 33
units on a scale
  Limbal study eye redness: Baseline: number analyzed (Participants) | 10 | 13 | 13
  Limbal study eye redness: Baseline | 0.608 (0.1919) | 0.615 (0.2379) | 0.625 (0.3917)
  Limbal study eye redness: Change at Week 12: number analyzed (Participants) | 9 | 13 | 12
  Limbal study eye redness: Change at Week 12 | 0.039 (0.0830) | 0.015 (0.1760) | 0.004 (0.2171)
  Limbal both eyes redness: Baseline: number analyzed (Participants) | 10 | 13 | 13
  Limbal both eyes redness: Baseline | 0.643 (0.2295) | 0.550 (0.1915) | 0.734 (0.3225)
  Limbal both eyes redness: Change at Week 12: number analyzed (Participants) | 9 | 13 | 12
  Limbal both eyes redness: Change at Week 12 | 0.038 (0.1413) | 0.031 (0.1473) | -0.050 (0.1340)
  Bulbar study eye redness: Baseline: number analyzed (Participants) | 10 | 13 | 13
  Bulbar study eye redness: Baseline | 0.975 (0.3482) | 1.062 (0.2807) | 0.965 (0.3132)
  Bulbar study eye redness: Change at Week 12: number analyzed (Participants) | 9 | 13 | 12
  Bulbar study eye redness: Change at Week 12 | 0.139 (0.2118) | -0.069 (0.3146) | -0.050 (0.3162)
  Bulbar both eyes redness: Baseline: number analyzed (Participants) | 10 | 13 | 13
  Bulbar both eyes redness: Baseline | 0.995 (0.3310) | 0.992 (0.2120) | 0.994 (0.2354)
  Bulbar both eyes redness: Change at Week 12: number analyzed (Participants) | 9 | 13 | 12
  Bulbar both eyes redness: Change at Week 12 | 0.064 (0.1949) | -0.038 (0.2444) | -0.089 (0.1939)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 13
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Lotemax Gel 0.5% and Restasis 0.05% | Lotemax Gel 0.5% | Restasis 0.05%
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/36 | 0/33
Other Adverse Events (participants affected / at risk) | 5/33 | 2/36 | 3/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lotemax Gel 0.5% and Restasis 0.05% (N=33) | Lotemax Gel 0.5% (N=36) | Restasis 0.05% (N=33)
Eye Irritation (Eye disorders) | 3 | 2 | 2
Eye Pruritus (Eye disorders) | 2 | 0 | 0
Instillation Site Pain (General disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.